CLINICAL TRIAL: NCT03780205
Title: Objective Adherence With Optical Correction in Children With Bilateral and Unilateral Refractive Amblyopia
Brief Title: Bilateral and Unilateral Amblyopia Treatment Study
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit sufficient number of subjects
Sponsor: Salus University (Other)
Responsible Party: Principal Investigator, Stanley Hatch, OD, MPH, Associate Professor, Salus University
Other Study IDs: HJWSH1810
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Amblyopia
Keywords: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bilateral Group: Patients have bilateral amblyopia, which is defined that best-corrected visual acuity of <20/30 each eye.
  Interventions: Other: Prescription glasses for bilateral amblyopia
- Unilateral Group: Patients have unilateral amblyopia, which is defined that best-corrected visual acuity of <20/30 in the amblyopic eye; and interocular difference of best-corrected visual acuity at least two logMAR lines.
  Interventions: Other: Prescription glasses for unilateral amblyopia

INTERVENTIONS:
Other: Prescription glasses for bilateral amblyopia — Correction of refractive error with prescription glasses both eyes
  Groups: Bilateral Group
Other: Prescription glasses for unilateral amblyopia — Correction of asymmetric refractive errors with lenses
  Groups: Unilateral Group

SUMMARY:
The purpose for this study is to investigate spectacle compliance and treatment outcome in bilateral and unilateral refractive amblyopia in children age 3 to <10 years old. Specifically, how frequently and for what duration is spectacle wear necessary to maximize best-corrected visual acuity by spectacle correction alone.

DETAILED DESCRIPTION:
The purpose for this study is to investigate spectacle compliance and treatment outcome in bilateral and unilateral refractive amblyopia in children age 3 to <10 years old. Specifically, how frequently and for what duration is spectacle wear necessary to maximize best-corrected visual acuity by spectacle correction alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to < 10 years
* Subjects and their parent/guardian speak and understand English adequately to complete the study protocol and give informed consent. Subjects have the ability to adhere to the study visit schedule.
* All refractive error measures below will be determined by cycloplegic retinoscopy by one of the study investigators during the comprehensive eye exam. Measures are in minus cylinder spectacle prescription format.

Inclusion criteria for bilateral amblyopia:

The major eligibility criteria include:

* Best-corrected visual acuity of <20/30 each eye.
* For hypermetropia:

  * Spherical equivalent >+2.00 D each eye.
  * Spherical equivalent difference between eyes <1.25 D.
* For astigmatism without hypermetropia criteria above or myopia criteria below:

  * >1.75 D each eye
  * Difference between eyes <1.25 D
* For myopia:

  * Spherical equivalent <-5.00.
  * Spherical equivalent difference between eyes <1.25 D.

Inclusion criteria for unilateral amblyopia:

The major eligibility criteria include:

* Presence of anisometropia or constant unilateral strabismus.
* Best-corrected visual acuity in the amblyopic eye <20/30; and interocular difference of best-corrected visual acuity at least two logMAR lines.
* For anisometropia:

  * Spherical equivalent ≥ 1.00 D interocular difference
  * Astigmatism >1.75 D interocular difference
* For constant unilateral strabismus where spectacle prescription is indicated. Examples where spectacle prescription is indicated include esotropia caused at least in part by an accommodative component or where significant refractive error in either eye warrants spectacle prescription for improved vision.

Exclusion Criteria:

* History of spectacle wear
* Previous treatment for amblyopia
* Active amblyopia treatment planned other than spectacles at enrollment
* Prior intraocular or refractive surgery
* Ocular or systemic abnormalities that the examining investigator deems could impact prognosis for visual improvement. Examples could include birth history that may have affected brain development, extremely low birth weight (<1.5 lbs), seizure disorders, cerebral palsy, optic nerve hypoplasia, cranial nerve palsy. Examples that would usually not exclude are off axis media opacity, low birth weight (2.0-3.5 lbs) without complication, mild limitation of extraocular muscle. Cognitive impairment that prohibits accurate data collection

Ages: 3 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Children age at 3 to < 10 years, who is newly diagnosed as amblyopia and prescribed with glasses.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
visual acuity change from the baseline | 8 weeks
  visual acuity change from the baseline in logMAR
adherence with optical treatment | 8 weeks
  The adherence recorded with the microsensor will be calculated as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hatch, OD, Principal Investigator — Salus University
Locations (1):
- Salus University, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided